CLINICAL TRIAL: NCT01052272
Title: Phase 2/3 Study of Effect of AT1RB Versus ACE Inhibitor in Addition to XO Inhibitor on Progression of LV Remodeling and Dysfunction in Diabetic Patients With Acute MI.
Brief Title: Impact of Diabetes on Left Ventricular Remodeling
Acronym: P3
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Dr. Louis J. Dell'Italia, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: F040105007
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes
Keywords: Diabetes; Acute MI; Ang II type-1 receptor blockade (AT1RB); LV remodeling; ACE inhibitor therapy; XO inhibitor, Allopurinol; Systolic dysfunction; Diastolic dysfunction; LV dimensions; Cardiac MRI
MeSH Terms: conditions — Diabetes Mellitus | interventions — Ramipril; candesartan cilexetil; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ramipril (Active Comparator): The starting dose of Ramipril will be 2.5 mg once daily and rapidly titrated upward to 5 mg once daily after 5 days if systolic blood pressure is greater than 100 mmHg. After one month the patient will return to clinic for blood pressure check and will be titrated up to 10 mg once daily.
  Interventions: Drug: Ramipril
- Candesartan cilexetil (Active Comparator): The starting dose of Candesartan cilexetil will be 4 mg or 8 mg once daily and doubled every 2 weeks, if systolic blood pressure is greater than 100 mmHg, to a maximum dose of 32 mg once daily. After one month the patient will return to clinic for blood pressure check and will be titrated up to 32 mg once daily.
  Interventions: Drug: Candesartan cilexetil
- Ramipril and Allopurinol (Active Comparator): The starting dose of Ramipril will be 2.5 mg once daily and rapidly titrated upward to 5 mg once daily after 5 days if systolic blood pressure is greater than 100 mmHg. After one month the patient will return to clinic for blood pressure check and will be titrated up to 10 mg once daily. It is anticipated that the starting dose of each drug will be initiated in hospital and that the second dose will be implemented prior to discharge from the hospital. The starting dose of Allopurinol is 300 mg daily.
  Interventions: Drug: Ramipril; Drug: Allopurinol
- Candesartan cilexetil and Allopurinol (Active Comparator): The starting dose of Candesartan cilexetil will be 4 mg or 8 mg once daily and doubled every 2 weeks, if systolic blood pressure is greater than 100 mmHg, to a maximum dose of 32 mg once daily. After one month the patient will return to clinic for blood pressure check and will be titrated up to 32 mg once daily. The starting dose of Allopurinol is 300 mg daily.
  Interventions: Drug: Candesartan cilexetil; Drug: Allopurinol

INTERVENTIONS:
Drug: Ramipril — The starting dose of Ramipril will be 2.5 mg once daily and rapidly titrated upward to 5 mg once daily after 5 days if systolic blood pressure is greater than 100 mmHg. After one month the patient will return to clinic for blood pressure check and will be titrated up to 10 mg once daily.
  Other Names: Altace
  Arms: Ramipril; Ramipril and Allopurinol
Drug: Candesartan cilexetil — The starting dose of Candesartan cilexetil will be 4 mg or 8 mg once daily and doubled every 2 weeks, if systolic blood pressure is greater than 100 mmHg, to a maximum dose of 32 mg once daily. After one month the patient will return to clinic for blood pressure check and will be titrated up to 32 mg once daily.
  Other Names: Atacand
  Arms: Candesartan cilexetil; Candesartan cilexetil and Allopurinol
Drug: Allopurinol — The starting dose of Allopurinol is 300 mg daily.
  Other Names: Altace
  Arms: Candesartan cilexetil and Allopurinol; Ramipril and Allopurinol

SUMMARY:
The investigators hypothesize that in patients with diabetes and acute myocardial infarction (MI), Ang II type-1 receptor blockade (AT1RB) attenuates left ventricle (LV) remodeling to a greater extent than angiotensin converting enzyme (ACE) inhibitor therapy and that the addition of xanthine oxidase (XO) inhibitor, Allopurinol, results in further improvement in LV remodeling and function in the follow-up phase after MI.

DETAILED DESCRIPTION:
Following myocardial infarction (MI), the incidence of heart failure and mortality rates are approximately two-fold higher in patients with diabetes compared to those without diabetes. This increased risk for heart failure and mortality appears to be refractory to currently available treatments such as angiotensin converting enzyme (ACE) inhibitors, despite the effectiveness of such treatments in reducing overall morbidity and mortality following MI. Hyperglycemia stimulates cardiomyocyte angiotensin II (Ang II) formation, which has been implicated in increased myocyte cell death in diabetes. Furthermore, in humans, chymase is the predominant pathway of Ang II formation and this pathway of Ang II production is not blocked by ACE inhibition. Therefore, in diabetes where Ang II levels may already be elevated due to hyperglycemia the increase in Ang II formation associated with left ventricular (LV) remodeling continued Ang II formation from chymase could be particularly detrimental.

In addition to enhanced Ang II production, hyperglycemia and diabetes also amplify the production of reactive oxygen species (ROS). ROS are associated with increased in LV remodeling and myocyte apoptosis. Furthermore, xanthine oxidase (XO), an important source of ROS in myocytes, is increased in a rat model of myocardial infarction and in diabetes. Thus, increased XO-mediated ROS production following MI may be especially damaging in diabetic patients where ROS production is already elevated. Interestingly, acute treatment with Allopurinol, an inhibitor of XO, improves cardiac function in heart failure and improves endothelial dysfunction in patients with type-2 diabetes.

To test our hypothesis the investigators will investigate the following aims in diabetic patients after acute MI:

Aim 1: Show that the progression of LV remodeling and dysfunction in diabetic patients will be attenuated to greater extent by AT1RB than by ACE inhibitor.

Aim 2: Show that the addition of XO inhibition results in further attenuation of LV remodeling than with AT1RB or ACE inhibitor alone.

Aim 3: Show that baseline and follow-up LV remodeling and dysfunction and inflammatory markers differ in diabetic and non-diabetic patients post-MI.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years old or older
2. MI documented by increase in troponin > 0.78 ng/ml or CKMB ≥ 3% of total CK

   Patients who have Type-2 diabetes defined by any one of the following:
3. Confirmed (i.e., two or more readings) fasting blood glucose >126mg/dl; or
4. Random glucose ≥200mg/dl; or
5. 2 hour glucose ≥200mg/dl following 75g of glucose; or
6. Current treatment with diet or oral agents directed at the control of hyperglycemia either alone or in combination with insulin; or
7. Current treatment with insulin with no prior history of diabetic ketoacidosis.

Exclusion Criteria:

1. Type-1 diabetes.
2. Class III or IV heart failure.
3. Cardiomyopathy (including hypertrophic and amyloidosis).
4. Congenital or pericardial diseases.
5. Intolerance to either ACE inhibitor, AT1-RB or allopurinol.
6. Renal failure with creatinine > 2.5 mg/dl.
7. Renal artery stenosis.
8. Severe comorbidity such as liver disease or malignancy.
9. Pregnancy (negative pregnancy test and effective contraceptive methods are required prior to enrollment of females of childbearing potential (not post-menopausal or surgically sterilized).
10. Chronic steroid use.
11. Unable to understand or cooperate with protocol requirements.
12. Severe claustrophobia.
13. Presence of a pacemaker or non-removable hearing aid.
14. Presence of metal clips in the body.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis J. Dell'Italia, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Background] Solomon SD, St John Sutton M, Lamas GA, Plappert T, Rouleau JL, Skali H, Moye L, Braunwald E, Pfeffer MA; Survival And Ventricular Enlargement (SAVE) Investigators. Ventricular remodeling does not accompany the development of heart failure in diabetic patients after myocardial infarction. Circulation. 2002 Sep 3;106(10):1251-5. doi: 10.1161/01.cir.0000032313.82552.e3. PMID 12208801
- [Background] Mukamal KJ, Nesto RW, Cohen MC, Muller JE, Maclure M, Sherwood JB, Mittleman MA. Impact of diabetes on long-term survival after acute myocardial infarction: comparability of risk with prior myocardial infarction. Diabetes Care. 2001 Aug;24(8):1422-7. doi: 10.2337/diacare.24.8.1422. PMID 11473080
- [Background] Melchior T, Kober L, Madsen CR, Seibaek M, Jensen GV, Hildebrandt P, Torp-Pedersen C. Accelerating impact of diabetes mellitus on mortality in the years following an acute myocardial infarction. TRACE Study Group. Trandolapril Cardiac Evaluation. Eur Heart J. 1999 Jul;20(13):973-8. doi: 10.1053/euhj.1999.1530. PMID 10361050
- [Background] Effect of ramipril on mortality and morbidity of survivors of acute myocardial infarction with clinical evidence of heart failure. The Acute Infarction Ramipril Efficacy (AIRE) Study Investigators. Lancet. 1993 Oct 2;342(8875):821-8. PMID 8104270
- [Background] Pfeffer MA, Braunwald E, Moye LA, Basta L, Brown EJ Jr, Cuddy TE, Davis BR, Geltman EM, Goldman S, Flaker GC, et al. Effect of captopril on mortality and morbidity in patients with left ventricular dysfunction after myocardial infarction. Results of the survival and ventricular enlargement trial. The SAVE Investigators. N Engl J Med. 1992 Sep 3;327(10):669-77. doi: 10.1056/NEJM199209033271001. PMID 1386652
- [Background] Fiordaliso F, Leri A, Cesselli D, Limana F, Safai B, Nadal-Ginard B, Anversa P, Kajstura J. Hyperglycemia activates p53 and p53-regulated genes leading to myocyte cell death. Diabetes. 2001 Oct;50(10):2363-75. doi: 10.2337/diabetes.50.10.2363. PMID 11574421
- [Background] Fiordaliso F, Li B, Latini R, Sonnenblick EH, Anversa P, Leri A, Kajstura J. Myocyte death in streptozotocin-induced diabetes in rats in angiotensin II- dependent. Lab Invest. 2000 Apr;80(4):513-27. doi: 10.1038/labinvest.3780057. PMID 10780668
- [Background] Urata H, Healy B, Stewart RW, Bumpus FM, Husain A. Angiotensin II-forming pathways in normal and failing human hearts. Circ Res. 1990 Apr;66(4):883-90. doi: 10.1161/01.res.66.4.883. PMID 2156635
- [Background] Brownlee M. Biochemistry and molecular cell biology of diabetic complications. Nature. 2001 Dec 13;414(6865):813-20. doi: 10.1038/414813a. PMID 11742414
- [Background] Giugliano D, Ceriello A, Paolisso G. Oxidative stress and diabetic vascular complications. Diabetes Care. 1996 Mar;19(3):257-67. doi: 10.2337/diacare.19.3.257. PMID 8742574
- [Background] Sorescu D, Griendling KK. Reactive oxygen species, mitochondria, and NAD(P)H oxidases in the development and progression of heart failure. Congest Heart Fail. 2002 May-Jun;8(3):132-40. doi: 10.1111/j.1527-5299.2002.00717.x. PMID 12045381
- [Background] Pimentel DR, Amin JK, Xiao L, Miller T, Viereck J, Oliver-Krasinski J, Baliga R, Wang J, Siwik DA, Singh K, Pagano P, Colucci WS, Sawyer DB. Reactive oxygen species mediate amplitude-dependent hypertrophic and apoptotic responses to mechanical stretch in cardiac myocytes. Circ Res. 2001 Aug 31;89(5):453-60. doi: 10.1161/hh1701.096615. PMID 11532907
- [Background] de Jong JW, Schoemaker RG, de Jonge R, Bernocchi P, Keijzer E, Harrison R, Sharma HS, Ceconi C. Enhanced expression and activity of xanthine oxidoreductase in the failing heart. J Mol Cell Cardiol. 2000 Nov;32(11):2083-9. doi: 10.1006/jmcc.2000.1240. PMID 11040111
- [Background] Matsumoto S, Koshiishi I, Inoguchi T, Nawata H, Utsumi H. Confirmation of superoxide generation via xanthine oxidase in streptozotocin-induced diabetic mice. Free Radic Res. 2003 Jul;37(7):767-72. doi: 10.1080/1071576031000107344. PMID 12911273
- [Background] Desco MC, Asensi M, Marquez R, Martinez-Valls J, Vento M, Pallardo FV, Sastre J, Vina J. Xanthine oxidase is involved in free radical production in type 1 diabetes: protection by allopurinol. Diabetes. 2002 Apr;51(4):1118-24. doi: 10.2337/diabetes.51.4.1118. PMID 11916934
- [Background] Cappola TP, Kass DA, Nelson GS, Berger RD, Rosas GO, Kobeissi ZA, Marban E, Hare JM. Allopurinol improves myocardial efficiency in patients with idiopathic dilated cardiomyopathy. Circulation. 2001 Nov 13;104(20):2407-11. doi: 10.1161/hc4501.098928. PMID 11705816
- [Background] Saavedra WF, Paolocci N, St John ME, Skaf MW, Stewart GC, Xie JS, Harrison RW, Zeichner J, Mudrick D, Marban E, Kass DA, Hare JM. Imbalance between xanthine oxidase and nitric oxide synthase signaling pathways underlies mechanoenergetic uncoupling in the failing heart. Circ Res. 2002 Feb 22;90(3):297-304. doi: 10.1161/hh0302.104531. PMID 11861418
- [Background] Butler R, Morris AD, Belch JJ, Hill A, Struthers AD. Allopurinol normalizes endothelial dysfunction in type 2 diabetics with mild hypertension. Hypertension. 2000 Mar;35(3):746-51. doi: 10.1161/01.hyp.35.3.746. PMID 10720589
- [Background] American Diabetes Association: clinical practice recommendations 1995. Diabetes Care. 1995 Jan;18 Suppl 1:1-96. No abstract available. PMID 7698058
- [Background] Diez J, Querejeta R, Lopez B, Gonzalez A, Larman M, Martinez Ubago JL. Losartan-dependent regression of myocardial fibrosis is associated with reduction of left ventricular chamber stiffness in hypertensive patients. Circulation. 2002 May 28;105(21):2512-7. doi: 10.1161/01.cir.0000017264.66561.3d. PMID 12034658
- [Background] Querejeta R, Varo N, Lopez B, Larman M, Artinano E, Etayo JC, Martinez Ubago JL, Gutierrez-Stampa M, Emparanza JI, Gil MJ, Monreal I, Mindan JP, Diez J. Serum carboxy-terminal propeptide of procollagen type I is a marker of myocardial fibrosis in hypertensive heart disease. Circulation. 2000 Apr 11;101(14):1729-35. doi: 10.1161/01.cir.101.14.1729. PMID 10758057
- [Background] Lopez B, Querejeta R, Varo N, Gonzalez A, Larman M, Martinez Ubago JL, Diez J. Usefulness of serum carboxy-terminal propeptide of procollagen type I in assessment of the cardioreparative ability of antihypertensive treatment in hypertensive patients. Circulation. 2001 Jul 17;104(3):286-91. doi: 10.1161/01.cir.104.3.286. PMID 11457746
- [Background] Cracowski JL, Tremel F, Marpeau C, Baguet JP, Stanke-Labesque F, Mallion JM, Bessard G. Increased formation of F(2)-isoprostanes in patients with severe heart failure. Heart. 2000 Oct;84(4):439-40. doi: 10.1136/heart.84.4.439. No abstract available. PMID 10995421
- [Background] Mallat Z, Philip I, Lebret M, Chatel D, Maclouf J, Tedgui A. Elevated levels of 8-iso-prostaglandin F2alpha in pericardial fluid of patients with heart failure: a potential role for in vivo oxidant stress in ventricular dilatation and progression to heart failure. Circulation. 1998 Apr 28;97(16):1536-9. doi: 10.1161/01.cir.97.16.1536. PMID 9593557
- [Background] Nonaka-Sarukawa M, Yamamoto K, Aoki H, Takano H, Katsuki T, Ikeda U, Shimada K. Increased urinary 15-F2t-isoprostane concentrations in patients with non-ischaemic congestive heart failure: a marker of oxidative stress. Heart. 2003 Aug;89(8):871-4. doi: 10.1136/heart.89.8.871. PMID 12860861
- [Background] Mak S, Newton GE. The oxidative stress hypothesis of congestive heart failure: radical thoughts. Chest. 2001 Dec;120(6):2035-46. doi: 10.1378/chest.120.6.2035. PMID 11742938
- [Background] Rouleau JL, Pitt B, Dhalla NS, Dhalla KS, Swedberg K, Hansen MS, Stanton E, Lapointe N, Packer M; Canadian Prospective RandOmized FlosequInan Longevity Evaluation Investigators. Prognostic importance of the oxidized product of catecholamines, adrenolutin, in patients with severe heart failure. Am Heart J. 2003 May;145(5):926-32. doi: 10.1016/s0002-8703(02)94782-4. PMID 12766756
- [Background] Lopez Farre A, Casado S. Heart failure, redox alterations, and endothelial dysfunction. Hypertension. 2001 Dec 1;38(6):1400-5. doi: 10.1161/hy1201.099612. PMID 11751725
- [Background] Heart Outcomes Prevention Evaluation Study Investigators; Yusuf S, Sleight P, Pogue J, Bosch J, Davies R, Dagenais G. Effects of an angiotensin-converting-enzyme inhibitor, ramipril, on cardiovascular events in high-risk patients. N Engl J Med. 2000 Jan 20;342(3):145-53. doi: 10.1056/NEJM200001203420301. PMID 10639539
- [Background] Pfeffer MA, Swedberg K, Granger CB, Held P, McMurray JJ, Michelson EL, Olofsson B, Ostergren J, Yusuf S, Pocock S; CHARM Investigators and Committees. Effects of candesartan on mortality and morbidity in patients with chronic heart failure: the CHARM-Overall programme. Lancet. 2003 Sep 6;362(9386):759-66. doi: 10.1016/s0140-6736(03)14282-1. PMID 13678868
- [Background] Granger CB, McMurray JJ, Yusuf S, Held P, Michelson EL, Olofsson B, Ostergren J, Pfeffer MA, Swedberg K; CHARM Investigators and Committees. Effects of candesartan in patients with chronic heart failure and reduced left-ventricular systolic function intolerant to angiotensin-converting-enzyme inhibitors: the CHARM-Alternative trial. Lancet. 2003 Sep 6;362(9386):772-6. doi: 10.1016/S0140-6736(03)14284-5. PMID 13678870
- [Background] Young JB, Dunlap ME, Pfeffer MA, Probstfield JL, Cohen-Solal A, Dietz R, Granger CB, Hradec J, Kuch J, McKelvie RS, McMurray JJ, Michelson EL, Olofsson B, Ostergren J, Held P, Solomon SD, Yusuf S, Swedberg K; Candesartan in Heart failure Assessment of Reduction in Mortality and morbidity (CHARM) Investigators and Committees. Mortality and morbidity reduction with Candesartan in patients with chronic heart failure and left ventricular systolic dysfunction: results of the CHARM low-left ventricular ejection fraction trials. Circulation. 2004 Oct 26;110(17):2618-26. doi: 10.1161/01.CIR.0000146819.43235.A9. Epub 2004 Oct 18. PMID 15492298
- [Background] Solomon SD, Wang D, Finn P, Skali H, Zornoff L, McMurray JJ, Swedberg K, Yusuf S, Granger CB, Michelson EL, Pocock S, Pfeffer MA. Effect of candesartan on cause-specific mortality in heart failure patients: the Candesartan in Heart failure Assessment of Reduction in Mortality and morbidity (CHARM) program. Circulation. 2004 Oct 12;110(15):2180-3. doi: 10.1161/01.CIR.0000144474.65922.AA. Epub 2004 Oct 4. PMID 15466644
- [Background] Wachtell K, Palmieri V, Olsen MH, Gerdts E, Papademetriou V, Nieminen MS, Smith G, Dahlof B, Aurigemma GP, Devereux RB. Change in systolic left ventricular performance after 3 years of antihypertensive treatment: the Losartan Intervention for Endpoint (LIFE) Study. Circulation. 2002 Jul 9;106(2):227-32. doi: 10.1161/01.cir.0000021601.49664.2a. PMID 12105163
- [Background] Rogers WJ, Bowlby LJ, Chandra NC, French WJ, Gore JM, Lambrew CT, Rubison RM, Tiefenbrunn AJ, Weaver WD. Treatment of myocardial infarction in the United States (1990 to 1993). Observations from the National Registry of Myocardial Infarction. Circulation. 1994 Oct;90(4):2103-14. doi: 10.1161/01.cir.90.4.2103. PMID 7923698
- [Background] Chandra NC, Ziegelstein RC, Rogers WJ, Tiefenbrunn AJ, Gore JM, French WJ, Rubison M. Observations of the treatment of women in the United States with myocardial infarction: a report from the National Registry of Myocardial Infarction-I. Arch Intern Med. 1998 May 11;158(9):981-8. doi: 10.1001/archinte.158.9.981. PMID 9588431
- [Background] Taylor HA Jr, Canto JG, Sanderson B, Rogers WJ, Hilbe J. Management and outcomes for black patients with acute myocardial infarction in the reperfusion era. National Registry of Myocardial Infarction 2 Investigators. Am J Cardiol. 1998 Nov 1;82(9):1019-23. doi: 10.1016/s0002-9149(98)00547-5. PMID 9817474
- [Background] Rogers WJ, Canto JG, Lambrew CT, Tiefenbrunn AJ, Kinkaid B, Shoultz DA, Frederick PD, Every N. Temporal trends in the treatment of over 1.5 million patients with myocardial infarction in the US from 1990 through 1999: the National Registry of Myocardial Infarction 1, 2 and 3. J Am Coll Cardiol. 2000 Dec;36(7):2056-63. doi: 10.1016/s0735-1097(00)00996-7. PMID 11127441
- [Background] Rogers WJ, Canto JG, Barron HV, Boscarino JA, Shoultz DA, Every NR. Treatment and outcome of myocardial infarction in hospitals with and without invasive capability. Investigators in the National Registry of Myocardial Infarction. J Am Coll Cardiol. 2000 Feb;35(2):371-9. doi: 10.1016/s0735-1097(99)00505-7. PMID 10676683

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ramipril | Candesartan Cilexetil | Ramipril and Allopurinol | Candesartan Cilexetil and Allopurinol
Started | 18 | 18 | 18 | 18
Completed | 13 | 11 | 10 | 11
Not Completed | 5 | 7 | 8 | 7
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — patient refuses follow-up | 5 | 4 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 2 | 3 | 2
Not completed — placed in long-term care | 0 | 0 | 1 | 0
Not completed — decline in health | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramipril | Candesartan Cilexetil | Ramipril and Allopurinol | Candesartan Cilexetil and Allopurinol | Total
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 11 | 10 | 45
  >=65 years | 6 | 6 | 7 | 8 | 27
Age Continuous [Mean (Standard Deviation); unit: years] | 58.17 (10.61) | 60.94 (11.27) | 60.67 (10.57) | 62 (10.86) | 60.44 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 8 | 3 | 16
  Male | 16 | 15 | 10 | 15 | 56
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 18 | 18 | 72

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular End Diastolic Volume Indexed to Body Surface Area (LVEDV/BSA)
Description: LVEDV/BSA: As an indicator of heart size, the blood volume of the heart is related to the body size. The relation of heart blood volume to body size is more accurate in determining pathology because larger people require a larger heart blood volume. The values that are too high or too low indicate a diseased myocardium. This is a measure of LV Diastolic Function. Since some visits did not occur at the scheduled 6 month intervals, the results have been divided into 3-month visit intervals.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Ramipril | Candesartan Cilexetil | Ramipril and Allopurinol | Candesartan Cilexetil and Allopurinol
Number analyzed (Participants) | 18 | 18 | 18 | 18
ml/m^2
  Month 0 (n=17,17,18,18) | 73.03 (20.34) | 78.06 (18.4) | 78.52 (19.31) | 79.03 (21.39)
  Month 6(n=14,11,11,12) | 74.10 (15.53) | 78.60 (24.30) | 86.13 (24.14) | 78.01 (14.49)
  Month 9(n=1,2,0,0) | 73.23 (NA) — n=1 | 93.57 (18.48) | NA (NA) — n=0 | NA (NA) — n=0
  Month12(n=12,11,11,11) | 75.34 (20.30) | 85.44 (20.87) | 83.95 (20.69) | 79.75 (19.9)
  Month 15(n=3,2,1,1) | 81.19 (5.96) | 90.20 (13.24) | 108.25 (NA) — n=1 | 63.1 (NA) — n=1
  Month 18(n=10,12,8,8) | 75.28 (14.48) | 82.74 (23.09) | 67.96 (12.86) | 84.95 (17.55)
  Month 21(n=3,0,0,1) | 71.99 (28.13) | NA (NA) — n=0 | NA (NA) — n=0 | 75.27 (NA) — n=1
  Month 24 (n=11,9,8,10) | 70.46 (17.17) | 84.28 (23.17) | 71.63 (8.59) | 79.72 (15.11)
  Month 27 (n=1,1,0,1) | 48.68 (NA) — n=1 | 76.65 (NA) — n=1 | NA (NA) — n=0 | 75.05 (NA) — n=1

2. Primary Outcome: Left Ventricular End-Diastolic Radius to Wall Thickness (LVED Radius/Wall Thickness)
Description: LVED Radius/Wall thickness As an indicator of heart muscle mass and heart volume chamber diameter, the end-diastolic radius indexed to end diastolic wall thickness determines whether there is an adequate amount of heart muscle to pump the heart blood volume obtained from a two-dimensional analysis. The values that are too high or too low indicate a diseased myocardium. This is a measure of LV Geometry. Since some visits did not occur at the scheduled 6 month intervals, the results have been divided into 3-month visit intervals for reporting purposes.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Ramipril | Candesartan Cilexetil | Ramipril and Allopurinol | Candesartan Cilexetil and Allopurinol
Number analyzed (Participants) | 18 | 18 | 18 | 18
unitless
  Month 0 (n=17,17,18,18) | 3.23 (0.77) | 3.14 (0.79) | 3.57 (0.98) | 3.45 (0.61)
  Month 6(n=14,11,11,12) | 3.32 (0.70) | 3.39 (0.44) | 4.04 (0.75) | 3.63 (0.61)
  Month 9(n=1,2,0,0) | 3.42 (NA) — n=1 | 4.14 (0.84) | NA (NA) — n=0 | NA (NA) — n=0
  Month 12(n=12,11,11,11) | 3.43 (0.71) | 3.68 (0.68) | 4.01 (0.71) | 3.42 (0.47)
  Month 15(n=3,2,1,1) | 3.44 (0.56) | 4.10 (1.10) | 4.57 (NA) — n=1 | 3.90 (NA) — n=1
  Month 18(n=10,12,8,8) | 3.60 (0.69) | 3.71 (0.76) | 3.60 (0.55) | 3.56 (0.48)
  Month 21(n=3,0,0,1) | 2.92 (0.43) | NA (NA) — n=0 | NA (NA) — n=0 | 4.24 (NA) — n=1
  Month 24 (n=11,9,8,10) | 3.46 (0.74) | 3.58 (0.69) | 3.61 (0.57) | 3.56 (0.37)
  Month 27 (n=1,1,0,1) | 3.12 (NA) — n=1 | 4.04 (NA) — n=1 | NA (NA) — n=0 | 4.29 (NA) — n=1

3. Primary Outcome: Left Ventricular End-diastolic Mass Indexed to Left Ventricular End-diastolic Volume (LVED Mass/LVEDV)
Description: LVED Mass/LVEDV: As an indicator of heart muscle mass and heart blood volume, the mass indexed to end diastolic volume determines whether there is an adequate amount of heart muscle to pump the heart blood volume obtained from a three-dimensional analysis. The values that are too high or too low indicate a diseased myocardium. This is a measure of LV Geometry. Since some visits did not occur at the scheduled 6 month intervals, the results have been divided into 3-month visit intervals for reporting purposes.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: g/ml
Arm/Group | Ramipril | Candesartan Cilexetil | Ramipril and Allopurinol | Candesartan Cilexetil and Allopurinol
Number analyzed (Participants) | 18 | 18 | 18 | 18
g/ml
  Month 0 (n=17,17,18,18) | 0.92 (0.25) | 0.95 (0.27) | 0.86 (0.26) | 0.87 (0.13)
  Month 6(n=14,11,11,12) | 0.87 (0.18) | 0.83 (0.13) | 0.71 (0.17) | 0.82 (0.12)
  Month 9(n=1,2,0,0) | 0.75 (NA) — n=1 | 0.67 (0.11) | NA (NA) — n=0 | NA (NA) — n=0
  Month 12(n=12,11,11,11) | 0.84 (0.18) | 0.78 (0.19) | 0.72 (0.15) | 0.86 (0.13)
  Month 15(n=3,2,1,1) | 0.81 (0.16) | 0.70 (0.18) | 0.57 (NA) — n=1 | 0.68 (NA) — n=1
  Month 18(n=10,12,8,8) | 0.79 (0.16) | 0.79 (0.22) | 0.83 (0.16) | 0.80 (0.12)
  Month 21(n=3,0,0,1) | 0.95 (0.25) | NA (NA) — n=0 | NA (NA) — n=0 | 0.69 (NA) — n=1
  Month 24 (n=11,9,8,10) | 0.84 (0.18) | 0.80 (0.20) | 0.80 (0.14) | 0.82 (0.08)
  Month 27 (n=1,1,0,1) | 0.93 (NA) — n=1 | 0.64 (NA) — n=1 | NA (NA) — n=0 | 0.69 (NA) — n=1

4. Primary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: LVEF is a calculation of heart pump function determined from the volume after complete filling minus the volume after complete contraction divided by the volume after complete filling. A value of 55% or greater is normal. This is a measure of LV Systolic Function. Since some visits did not occur at the scheduled 6 month intervals, the results have been divided into 3-month visit intervals for reporting purposes
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Ramipril | Candesartan Cilexetil | Ramipril and Allopurinol | Candesartan Cilexetil and Allopurinol
Number analyzed (Participants) | 18 | 18 | 18 | 18
percent
  Month 0 (n=17,17,18,18) | 52.19 (10.65) | 56.36 (12.34) | 53.37 (10.01) | 52.68 (13.90)
  Month 6(n=14,11,11,12) | 54.20 (10.27) | 56.82 (10.81) | 52.80 (15.66) | 57.28 (9.17)
  Month 9(n=1,2,0,0) | 64.98 (NA) — n=1 | 42.62 (1.95) | NA (NA) — n=0 | NA (NA) — n=0
  Month 12(n=12,11,11,11) | 52.76 (9.94) | 52.37 (11.41) | 51.74 (15.54) | 56.11 (11.33)
  Month 15(n=3,2,1,1) | 52.13 (14.08) | 39.88 (2.76) | 34.89 (NA) — n=1 | 54.46 (NA) — n=1
  Month 18(n=10,12,8,8) | 55.02 (13.24) | 56.33 (10.26) | 54.05 (9.96) | 57.82 (10.97)
  Month 21(n=3,0,0,1) | 51.27 (1.73) | NA (NA) — n=0 | NA (NA) — n=0 | 56.17 (NA) — n=1
  Month 24 (n=11,9,8,10) | 57.18 (9.79) | 51.70 (10.02) | 55.59 (9.47) | 55.79 (10.53)
  Month 27 (n=1,1,0,1) | 50.73 (NA) — n=1 | 54.17 (NA) — n=1 | NA (NA) — n=0 | 54.40 (NA) — n=1

5. Primary Outcome: Left Ventricular End Systolic Volume Indexed to Body Surface Area (LVESV/BSA)
Description: LVESV/BSA: The end systolic volume is the blood volume of the heart at the end of contraction and is an index of the pump function of the heart. This relation to body size is more accurate in determining pathology because larger people require a larger heart blood volume. The values that are too high or too low indicate a diseased myocardium. This is a measure of LV Systolic Function. Since some visits did not occur at the scheduled 6 month intervals, the results have been divided into 3-month visit intervals.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: ml/m^2
Arm/Group | Ramipril | Candesartan Cilexetil | Ramipril and Allopurinol | Candesartan Cilexetil and Allopurinol
Number analyzed (Participants) | 18 | 18 | 18 | 18
ml/m^2
  Month 0 (n=17,17,18,18) | 36.20 (16.64) | 35.26 (16.08) | 37.91 (16.63) | 39.49 (21.97)
  Month 6(n=14,11,11,12) | 34.77 (13.56) | 35.26 (18.36) | 42.88 (25.33) | 34.15 (12.80)
  Month 9(n=1,2,0,0) | 25.64 (NA) — n=1 | 53.87 (12.43) | NA (NA) — n=0 | NA (NA) — n=0
  Month 12(n=12,11,11,11) | 36.82 (15.88) | 42.27 (19.83) | 42.34 (25.18) | 36.07 (16.24)
  Month 15(n=3,2,1,1) | 39.42 (14.05) | 54.04 (5.47) | 70.48 (NA) — n=1 | 28.74 (NA) — n=1
  Month 18(n=10,12,8,8) | 35.30 (17.21) | 37.76 (18.48) | 30.39 (4.61) | 37.18 (15.95)
  Month 21(n=3,0,0,1) | 35.23 (14.52) | NA (NA) — n=0 | NA (NA) — n=0 | 32.99 (NA) — n=1
  Month 24 (n=11,9,8,10) | 31.17 (14.47) | 41.72 (18.48) | 31.56 (6.52) | 35.99 (13.65)
  Month 27 (n=1,1,0,1) | 23.98 (NA) — n=1 | 35.13 (NA) — n=1 | NA (NA) — n=0 | 34.22 (NA) — n=1

6. Primary Outcome: LV End Systolic Maximum Shortening (LVES Max Shortening)
Description: By identifying three points in three different planes in the heart muscle, the maximum shortening is the average of the difference between the distance between these three points at the end of filling of the heart and the end of contraction divided by the length at the end of filling times 100. The maximum shortening is a three dimensional analysis. The higher values indicate a healthy heart. This is a measure of LV Systolic Function. Since some visits did not occur at the scheduled 6 month intervals, the results have been divided into 3-month visit intervals for reporting purposes.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: percent of length at end of filling
Arm/Group | Ramipril | Candesartan Cilexetil | Ramipril and Allopurinol | Candesartan Cilexetil and Allopurinol
Number analyzed (Participants) | 18 | 18 | 18 | 18
percent of length at end of filling
  Month 0 (n=17,17,17,18) | 15.81 (3.56) | 16.68 (3.12) | 15.84 (2.70) | 16.00 (2.77)
  Month 6(n=14,11,10,12) | 16.88 (1.90) | 17.50 (2.07) | 18.72 (2.4) | 18.50 (2.0)
  Month 9(n=1,2,0,0) | 18.43 (NA) — n=1 | 19.08 (2.78) | NA (NA) — n=0 | NA (NA) — n=0
  Month 12(n=11,11,10,10) | 14.57 (2.91) | 17.13 (1.94) | 17.96 (1.68) | 18.51 (2.41)
  Month 15(n=3,2,1,1) | 17.06 (1.83) | 16.28 (2.42) | 14.22 (NA) — n=1 | 16.36 (NA) — n=1
  Month 18(n=10,12,7,8) | 17.26 (1.46) | 17.55 (1.62) | 17.46 (1.19) | 17.52 (1.6)
  Month 21(n=3,0,0,1) | 16.68 (1.27) | NA (NA) — n=0 | NA (NA) — n=0 | 17.89 (NA) — n=1
  Month 24 (n=11,9,8,10) | 15.67 (3.36) | 16.62 (1.32) | 17.52 (1.17) | 17.85 (1.37)
  Month 27 (n=1,1,0,1) | 13.70 (NA) — n=1 | 20.38 (NA) — n=0 | NA (NA) — n=0 | 16.59 (NA) — n=1

7. Primary Outcome: Peak Early Filling Rate Normalized to EDV
Description: The Peak Early Filling Rate Normalized to EDV is calculated from the slope of the volume during the early filling of the heart with respect to time. The higher values indicate a very healthy heart muscle and lower values are indicative of a very stiff muscle. This is a measure of LV Diastolic Function. Since some visits did not occur at the scheduled 6 month intervals, the results have been divided into 3-month visit intervals for reporting purposes.
Time Frame: 5 visits per Participant over 2 years (about every 6 months)
Population: intent to treat
Measure: Mean (Standard Deviation); unit: 1/sec
Arm/Group | Ramipril | Candesartan Cilexetil | Ramipril and Allopurinol | Candesartan Cilexetil and Allopurinol
Number analyzed (Participants) | 18 | 18 | 18 | 18
1/sec
  Month 0 (n=17,17,18,18) | 1.93 (0.69) | 2.01 (0.76) | 2.11 (0.56) | 2.0 (0.74)
  Month 6(n=14,11,11,12) | 1.74 (0.77) | 2.02 (0.81) | 2.03 (0.95) | 1.98 (0.73)
  Month 9(n=1,2,0,0) | 2.50 (NA) — n=1 | 1.13 (0.83) | NA (NA) — n=0 | NA (NA) — n=0
  Month 12(n=12,11,11,11) | 1.80 (0.60) | 1.90 (0.71) | 1.93 (0.45) | 1.77 (0.83)
  Month 15(n=3,2,1,1) | 2.02 (1.09) | 1.48 (0.58) | 1.56 (NA) — n=1 | 2.28 (NA) — n=1
  Month 18(n=10,12,8,8) | 1.91 (0.52) | 1.93 (0.84) | 1.89 (0.78) | 2.05 (0.59)
  Month 21(n=3,0,0,1) | 1.69 (0.42) | NA (NA) — n=0 | NA (NA) — n=0 | 2.50 (NA) — n=1
  Month 24 (n=11,9,8,10) | 2.05 (0.81) | 1.65 (0.55) | 1.88 (0.50) | 1.82 (0.78)
  Month 27 (n=1,1,0,1) | 1.34 (NA) — n=1 | 1.10 (NA) — n=1 | NA (NA) — n=0 | 2.15 (NA) — n=1

ADVERSE EVENTS:
Arm/Group | Ramipril | Candesartan Cilexetil | Ramipril and Allopurinol | Candesartan Cilexetil and Allopurinol
Serious Adverse Events (participants affected / at risk) | 4/18 | 6/18 | 9/18 | 5/18
Other Adverse Events (participants affected / at risk) | 3/18 | 4/18 | 6/18 | 3/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Ramipril (N=18) | Candesartan Cilexetil (N=18) | Ramipril and Allopurinol (N=18) | Candesartan Cilexetil and Allopurinol (N=18)
cardiac catheterization performed (Cardiac disorders) | 1/17 (1) | 0 (0) | 1 (1) | 1 (1)
left above-knee amputation related to occlusion of his left external iliac artery (Vascular disorders) | 1/17 (1) | 0 (0) | 0 (0) | 0 (0)
coronary artery bypass grafting (Cardiac disorders) | 1/17 (1) | 2 (2) | 0 (0) | 1 (1)
hospitalized for chest pain; no surgical intervention (Cardiac disorders) | 1/17 (1) | 2 (2) | 0 (0) | 0 (0)
hospitalized for elective abdominal aortogram (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hospitalized for a critically high PT/INR (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hospitalized due to chest pain; depressed TSH of 0.009 and hematocrit of 22 with a negative hemocult (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hospitalized for prophylactic ICD implantation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
death due to cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
chronic anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hospitalized --paroxysmal atrial fibrillation, acute gouty arthritis, chronic renal failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hospitalized for anterior cervical discectomy of C5-C6 (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hospitalized for hematuria brought on by cystoscopy and right ureteroscopy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hospitalized for pneumonia and acute exudative tonsillitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hospitalized for acute pyelonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hospitalized for fever, cough, and general malaise; Hemodialysis was performed twice (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
infection resulting to altered mental status; episode of major depression; renal failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
death due to heart failure and renal failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
adenocarcinoma of the pancreas (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
elevated WBC; Chest x-ray revealed pleural thickening; cultures revealed klebsiella oxytoca (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
acute anterior left middle cerebral artery distribution infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
aortic valve replacement (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
coronary artery stent (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
enterococcus endocarditis; ischemic right leg and GI bleed. (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
adenosine MIBI GXT positive for ischemic heart disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
coronary angioplasty (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
episode of slurred speech and memory loss at home (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramipril (N=18) | Candesartan Cilexetil (N=18) | Ramipril and Allopurinol (N=18) | Candesartan Cilexetil and Allopurinol (N=18)
WORSENING RIGHT HIP (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
worsening lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
abdominal cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
increased shortness of breath (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STERNOTOMY MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE RENAL INSUFFICIENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHEST WALL PAIN (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BILATERAL HIP ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INTOLERANCE TO ACE-I (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GOUT (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CATARACT REPAIR LEFT EYE (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOWER PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERKALEMIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SEVERE AORTIC REGURGITATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
placement of AV fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No